CLINICAL TRIAL: NCT01174095
Title: A Post Ten Year Follow up Assessment of a Phase I Trial of Angiogenic Gene Therapy for the Treatment of Coronary Artery Disease Using Direct Intramyocardial Administration of an Adenovirus Vector Expressing the VEGF121 cDNA
Brief Title: Post Ten Year Follow up Assessment of a Phase I Trial of Angiogenic Gene Therapy
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Stony Brook University (Other)
Responsible Party: Sponsor
Other Study IDs: 0905010396
Record Dates: First submitted 2010-07-30; First posted 2010-08-03 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Coronary Artery Disease; Ischemia
Keywords: Diffuse Coronary Artery Disease; Ischemic Myocardium; Ischemia
MeSH Terms: conditions — Coronary Artery Disease; Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Follow-up Group: Subjects who received AdGVVEGF121cDNA in either IRB protocol #0794-894 entitled "Phase I Study of Direct Administration of a Replication Deficient Adenovirus Vector (AdGVVEGF121.10) Containing the VEGF121 cDNA to the Ischemic Myocardium of Individuals with Diffuse Coronary Artery Disease" or IRB protocol #0297-693 entitled "Phase I Study of Direct Administration of a Replication Deficient Adenovirus Vector (AdGVVEGF121.10) Containing the VEGF121 cDNA to the Ischemic Myocardium of Individuals with Diffuse Coronary Artery Disease Via Minimally Invasive Surgery".

SUMMARY:
The primary aim of the study is to assess and follow-up subjects that received AdGVVEGF121cDNA in IRB protocol #0794-894 entitled "Phase I Study of Direct Administration of a Replication Deficient Adenovirus Vector (AdGVVEGF121.10) Containing the VEGF121 cDNA to the Ischemic Myocardium of Individuals with Diffuse Coronary Artery Disease" and IRB protocol #0297-693 entitled "Phase I Study of Direct Administration of a Replication Deficient Adenovirus Vector (AdGVVEGF121.10) Containing the VEGF121 cDNA to the Ischemic Myocardium of Individuals with Diffuse Coronary Artery Disease Via Minimally Invasive Surgery".

DETAILED DESCRIPTION:
A research coordinator from Weill Cornell Medical College will survey the medical records of all 31 subjects, and obtain contact information for all living subjects. Living subjects will be called by the research coordinator at Stony Brook University Medical Center and invited to participate in the current follow-up study, which will entail a full medical chart review. If the potential subject is interested, he/she will be invited to Stony Brook University Medical Center where Dr. Rosengart or a designated co-investigator conducts the informed consent process. However, subjects who are unable to travel to Stony Brook University Medical Center will be mailed the consent form. Those who consent to participate will compile their medical records and send them to Stony Brook University Medical Center. The research coordinator at Stony Brook will conduct a chart review in order to collect information regarding the subject's medication, evaluation and surgical history over the past 10 years. This information will include cardiac health evaluations such as 99mTc-sestamibi SPECT, treadmill exercise tolerance test and cardiac specific blood tests. These parameters will be compared to evaluations done at baseline and evaluations done at the subject's last visit as a participant of either Institutional Review Board (IRB) protocol #0794-894 or #0297-693.

ELIGIBILITY:
Inclusion Criteria:

* Subjects for this study will be recruited from the population of subjects who participated in 2 previous Weill Cornell Medical College IRB gene transfer studies using AdGVVEGF121.10:

  1. IRB protocol #0794-894 entitled "Phase I Study of Direct Administration of a Replication Deficient Adenovirus Vector (AdGVVEGF121.10) Containing the VEGF121 cDNA to the Ischemic Myocardium of Individuals with Diffuse Coronary Artery Disease" and
  2. IRB protocol #0297-693 entitled "Phase I Study of Direct Administration of a Replication Deficient Adenovirus Vector (AdGVVEGF121.10) Containing the VEGF121 cDNA to the Ischemic Myocardium of Individuals with Diffuse Coronary Artery Disease Via Minimally Invasive Surgery."

Exclusion Criteria:

* Subjects for this study will be recruited from the population of subjects who participated in 2 previous Weill Cornell Medical College IRB gene transfer studies using AdGVVEGF121.10:

  1. IRB protocol #0794-894 entitled "Phase I Study of Direct Administration of a Replication Deficient Adenovirus Vector (AdGVVEGF121.10) Containing the VEGF121 cDNA to the Ischemic Myocardium of Individuals with Diffuse Coronary Artery Disease" and
  2. IRB protocol #0297-693 entitled "Phase I Study of Direct Administration of a Replication Deficient Adenovirus Vector (AdGVVEGF121.10) Containing the VEGF121 cDNA to the Ischemic Myocardium of Individuals with Diffuse Coronary Artery Disease Via Minimally Invasive Surgery."

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These subjects have clinically significant coronary artery disease (CAD) and have received direct myocardial injection of AdGVVEGF121.10 expressing the human vascular endothelial growth factor (VEGF) 121 cDNA to induce therapeutic angiogenesis.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2009-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Canadian Cardiovascular Society Angina Score | 10 Years
  The Canadian Cardiovascular Society Angina Score will be graded as:
  Grade I Stable angina develops upon strenuous, rapid, and/or prolonged exertion during work or recreation but is not induced by ordinary physical activity..
  Grade II
  Stable angina is characterized by a slight limitation of ordinary activity and is induced by:
  Walking uphill or climbing stairs rapidly Walking or stair-climbing after meals Walking more than two level blocks or climbing more than one flight of ordinary stairs at a normal pace and in normal conditions Emotional stress During the few hours after waking
  Grade III Stable angina is characterized by marked limitation of ordinary physical activity. It is induced by walking one or two level blocks and climbing one flight of stairs in normal conditions and at a normal pace.
  Grade IV Stable angina is characterized by an inability to carry on any physical activity without discomfort. Angina syndrome may be present at rest.

SECONDARY OUTCOMES:
Survival Rate | 10 Years
  It is the percentage of people in the study that are still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Weill Cornell Medicine, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York

IPD SHARING:
Plan to Share IPD: Undecided